CLINICAL TRIAL: NCT00681005
Title: A Comparative Study of Proton-pump Inhibitor Tests for Chinese Reflux Patients in Relation to the CYP2C19 Genotypes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 950204
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: GERD
Keywords: PPI test; gastroesophageal reflux disease; CYP2C19; rabeprazole; pantoprazole
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Rabeprazole; Pantoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rabeprazole (Active Comparator): Rabeprazole 1 # qd
  Interventions: Drug: rabeprazole
- pantoprazole (Active Comparator): Pantoprazole 1# qd
  Interventions: Drug: pantoprazole

INTERVENTIONS:
Drug: rabeprazole — 20 mg bid for 14 days
  Other Names: Pariet
  Arms: Rabeprazole
Drug: pantoprazole — pantoprazole 40 mg bid
  Other Names: Pantoloc
  Arms: pantoprazole

SUMMARY:
Backgrounds & Aims: Proton-pump inhibitor (PPI) test has been proposed as a valuable tool in the diagnosis of gastroesophageal reflux disease (GERD) in Western populations. We assumed that a higher prevalence of poor metabolizers in Chinese population might affect the diagnostic accuracy of a PPI test.

Methods: In this open-label, randomized trial, patients with symptoms suggestive of GERD were randomly assigned to receive a 2-week test with daily rabeprazole 40-mg or daily pantoprazole 80-mg after diagnostic endoscopy. Therapeutic response was assessed with a five-grade daily record. Genotypes of cytochrome P450 (CYP) 2C19 polymorphism were determined.

DETAILED DESCRIPTION:
As described above

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with symptoms suggesting GERD will be enrolled from gastroenterology outpatient clinics in our academic institute. The typical GERD symptom was defined as heartburn and/or regurgitation at least 3 episodes per week in recent 3 months.

Exclusion Criteria:

* Those who were under maintenance PPI treatment, have a medical contraindication to PPI therapy, report a history of peptic ulcer disease or gastrointestinal surgery, malignancy proven by endoscopy, or unwilling or unable to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2006-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
at least 50% reduction of symptoms | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, MD, PhD, Study Director — National Taiwan University Hospital